CLINICAL TRIAL: NCT07215494
Title: A Clinical Study on Minimal Residual Disease in Patients With Systemic Light Chain Amyloidosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujun DONG, chief of department of hematology, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUFH202510
Record Dates: First submitted 2025-10-02; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Light Chain (AL) Amyloidosis; MRD
Keywords: light chain amyloidosis; MRD; ASCT
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First-Line Treatment for MRD-Positive Patients Undergoing ASCT (Experimental): First-Line treatment with Dara-CyBorD achieves CR, but MRD-Positive patients are recommended to undergo ASCT.
  Interventions: Drug: First-Line Dara-BorCyD Treatment

INTERVENTIONS:
Drug: First-Line Dara-BorCyD Treatment — First-Line Dara-BorCyD Treatment Achieves CR, but ASCT is Recommended for MRD-Positive Patients

SUMMARY:
Before effective treatment, the prognosis of patients with AL amyloidosis is very poor, with a median survival of approximately 12 months. In recent decades, with the development of new drugs, the treatment paradigm for AL amyloidosis has undergone significant changes, and the prognosis has improved dramatically. Achieving very good partial response (VGPR) or even complete response (CR) can lead to higher organ response and longer survival. However, not all patients who achieve ≥VGPR reach organ response, which may be related to the presence of small residual plasma cell clones in these patients. The ongoing production of monoclonal light chains deposits into tissues and organs, causing continuous damage, making organ response difficult. With the development of new drugs, the rate of hematologic CR has continuously increased, and the advancement of minimal residual disease (MRD) detection technologies in recent years has led to increasing attention to MRD in AL amyloidosis research. Therefore, in this era of advancing new drugs, MRD negativity may become a higher clinical treatment goal for AL amyloidosis, further improving long-term prognosis for patients.

Our department plans to conduct a single-center, prospective clinical study aimed at exploring the MRD status in patients who achieve hematologic CR after first-line induction chemotherapy (Dara-CyBorD), and further investigating whether autologous stem cell transplantation in MRD-positive CR patients who meet transplant criteria can further improve organ response, progression-free survival, and overall survival.

DETAILED DESCRIPTION:
Light chain amyloidosis (AL amyloidosis), as a plasma cell disorder, is caused by a typically small and slowly proliferating clone of plasma cells in the bone marrow. The light chains produced by this clone misfold, forming amyloid fibrils that deposit in various tissues and organs, leading to progressive organ dysfunction. Prior to effective treatment, the prognosis for AL amyloidosis patients is very poor, with a median survival of approximately 12 months. In recent decades, with continuous improvements in patient selection criteria for autologous hematopoietic stem cell transplantation (ASCT) and the development of novel drugs such as proteasome inhibitors, the treatment landscape for AL amyloidosis has changed significantly, resulting in a marked improvement in patient prognosis.

Hematologic response assessment is a primary focus during treatment, with achieving very good partial response (VGPR) or even complete response (CR) leading to higher rates of organ response and longer survival. However, not all patients who achieve ≥VGPR reach organ response. This may be due to the presence of minimal residual plasma cell clones, which continue to produce monoclonal light chains that deposit in tissues and organs, causing ongoing damage, making organ response difficult. With the continuous development of novel drugs, the rate of hematologic CR has improved, and recent advancements in minimal residual disease (MRD) detection techniques, have increasingly drawn attention in AL amyloidosis research. Therefore, in an era of continuous drug development, achieving MRD negativity may become an important clinical treatment goal for AL amyloidosis, further improving long-term patient prognosis.

A favorable result from the 2021 randomized clinical trial (NCT03201965) led to the Dara-CyBorD regimen becoming the first FDA-approved first-line treatment in Europe and the U.S., which has sparked some debate about the role of ASCT. Dara can lead to early and deep hematologic remission, with a CR rate comparable to ASCT. Some studies have shown that patients receiving ASCT as first-line treatment have higher MRD-negative rates compared to those undergoing chemotherapy alone. MRD negativity is associated with better organ response and longer survival. However, there is currently no data comparing the MRD-negative rates between Dara and ASCT. ASCT can provide early and deep hematologic remission, and more importantly, long-lasting deep remission. Studies show that the median duration of hematologic CR in ASCT patients is 12.3 years, with 45% of patients remaining relapse-free 15 years after transplantation. In contrast, there is no data available on the duration of deep remission with Dara. In conclusion, for patients with AL amyloidosis who meet the ASCT criteria, ASCT may still be the preferred treatment.

Based on the favorable results of MRD in AL amyloidosis research and the continued advantages of ASCT (autologous stem cell transplantation) in the era of Dara, our department plans to conduct a single-center, prospective clinical study. The main objective of the study is to explore the MRD status in patients who achieve hematologic CR (complete response) after first-line induction chemotherapy (Dara-CyBorD). Additionally, the study will investigate whether ASCT in MRD-positive CR patients who meet transplantation criteria can further improve organ response, progression-free survival, and overall survival. Through MRD detection, this study aims to achieve deeper hematologic remission in the era of novel drugs, ultimately improving the long-term prognosis of AL amyloidosis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-70 years (inclusive), no gender restriction;
2. Newly diagnosed AL amyloidosis patients;
3. Meet ASCT eligibility criteria and have a willingness to undergo ASCT;
4. Achieved hematological complete response (CR) after 2-4 cycles of Dara-CyBorD induction chemotherapy.

Exclusion Criteria:

1. Secondary to multiple myeloma or lymphoplasmacytic lymphoma, such as Waldenström's macroglobulinemia;
2. Co-existing other active malignant tumors;
3. Co-existing other systemic diseases deemed unsuitable for inclusion by the investigator, such as newly developed severe cardiovascular and cerebrovascular diseases, or severe infections.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Organ Response Rates | 2 years
Progression-Free Survival | 2 years
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided